CLINICAL TRIAL: NCT01582815
Title: A Multicenter, Double-Blind, Placebo-Controlled Study of JNJ-40411813 as Adjunctive Treatment to an Antidepressant in Adults With Major Depressive Disorder With Anxiety Symptoms
Brief Title: A Study of JNJ-40411813 as Supplementary Treatment to an Antidepressant in Adults With Depression and Anxiety Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100851; 40411813DAX2001 (Other: Janssen Research & Development, LLC); 2011-006121-26 (EudraCT Number)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Anxiety symptoms; JNJ-40411813
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders | interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-40411813 (Experimental)
  Interventions: Drug: JNJ-40411813
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-40411813 — Type= range, unit= mg, number= 25 to 150, form= capsules, route= oral administration. JNJ-40411813 will be administered twice daily during 8 weeks, following fixed and flexible schedules in which the dose can range from 25 mg to 150 mg.
  Arms: JNJ-40411813
Drug: Placebo — Form= capsule, route= oral administration. Matching placebo will be administered twice daily during 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and overall safety and tolerability of treatment with adjunctive JNJ-40411813 compared to placebo in patients with MDD with anxiety symptoms being treated with an antidepressant.

DETAILED DESCRIPTION:
This is a multicenter, double-blind (neither physician nor patient knows the treatment that the patient receives), placebo-controlled study in adult patients with Major Depressive Disorder (MDD) with anxiety symptoms of relevant severity. The study will consist of 3 phases: a screening phase of up to 2 weeks, an 8-week double-blind treatment phase, and a 2-week post-treatment (follow up) phase. Patients will continue to take the same daily dose of their antidepressant (as directed by the investigator) at the same time of day, from screening through the end of the study, including the post-treatment phase. The total study duration for each patient will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD); patients with a diagnosis of comorbid Generalized Anxiety Disorder, Social Anxiety Disorder, or Panic Disorder may be included, if the investigator considers MDD to be the primary diagnosis
* A 17-item Hamilton Depression Rating Scale (HDRS17) total score =>18
* A HDRS17 anxiety/somatization factor score =>7
* Is receiving an antidepressant

Exclusion Criteria:

* Has other psychiatric condition, including, but not limited to, MDD with psychotic features, bipolar disorder, obsessive-compulsive disorder, post-traumatic stress disorder, borderline personality disorder, eating disorder, or schizophrenia
* Has a length of current Major Depressive Episode (MDE) >6 months
* Has a current or recent history of clinically significant suicidal ideation within the past 6 months, or a history of suicidal behavior within the past year
* Not including the inadequate response to the current antidepressant, has more than 1 failed antidepressant treatment of adequate dose and duration in the current MDE

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The change from baseline to endpoint on the Hamilton Anxiety Rating scale (HAM-A6) score | Baseline, Week 4
  The HAM-A6 is a 6-item subscale derived from the original Hamilton Anxiety scale (HAM-A). The rating scale measures the severity of anxiety symptomatology. Higher scores represent more severe anxiety symptoms.

SECONDARY OUTCOMES:
The change from baseline to endpoint on the Hamilton Depression Rating Scale (HDRS17) total score | Baseline, Week 4
  The HDRS17 is a clinician-administered rating scale designed to assess the severity of symptoms in patients diagnosed with depression with a score range of 0 to 52. Questions are related to symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss. The higher the score, the more severe the depression.
The change from baseline to endpoint on the SIGH-A (Structured Interview Guide of the Hamilton Anxiety Scale 14-item HAM-A) total score | Baseline, Week 4
  The (HAM-A) is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. The answers range from 0 which signifies a complete lack of that symptom to 4, which indicates a very severe show of anxiety with that symptom.
The change from baseline to endpoint in the Clinical Global Impression - Improvement (CGI-I) scale | Baseline, Week 4
  The CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
The change from baseline to endpoint in the Hamilton Depression Rating Scale (HDRS17) anxiety/somatization factor total score | Baseline, Week 4
  The HDRS17 is a clinician-administered rating scale designed to assess the severity of symptoms in patients diagnosed with depression with a score range of 0 to 52. Questions are related to symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss. The higher the score, the more severe the depression.
The change from baseline to endpoint in the HAM-D6 score | Baseline, Week 4
  The HAM-D6 is a 6-item subscale derived from the Hamilton Depression Rating Scale (HDRS17). The rating scale measures the severity of depressive symptomatology. Higher scores represent more severe depressive symptoms.
The change from baseline to endpoint in the Inventory of Depressive Symptomatolgy -Clinician rated (IDS-C30) total score | Baseline, Week 6
  The IDS-C30 is a clinician administered 30 item depression specific severity rating scale designed to measure specific signs and symptoms of depression including melancholic, atypical and anxious features. Scores range from 0 to 84 with higher scores representing greater severity of depressive symptoms.
The change from baseline to endpoint in the Inventory of Depressive Symptomatology - Clinician-Rated (IDS-C30) anxiety subscale | Baseline, Week 4
  The IDS-C30 is a clinician administered 30 item depression specific severity rating scale designed to measure specific signs and symptoms of depression including melancholic, atypical and anxious features. The anxiety subscale includes five anxiety symptoms: anxious mood, somatic complaints, sympathetic arousal, panic, and gastrointestinal symptoms. The rating scale measures the severity of anxiety symptomatology. Higher scores represent more severe anxiety symptoms.
The change from baseline to Week 4 in the Work Limitations Questionnaire (WLQ) | Baseline, Week 4
  The WLQ is a 25-item questionnaire self-report rating scale developed to measure the on-the-job impact of chronic health problems and/or treatment ("work limitations"), with a recall period of the previous 2 weeks. It comprises four dimensions of limitations: handling time, physical, mental-interpersonal, and output demands. Patients respond to each item with options ranging from "Almost all of the time" to "none of the time", or "Does not apply to my job". The global score ranges from 0 to 100 with lower score indicating low level of work limitations.
The change from baseline to endpoint on the Perceived Stress Scale (PSS) | Baseline, Week 4
  The PSS is a 10-item, self-reported unidimensional instrument developed to measure perceived stress in response to situations in a person's life. Prevalence of an item within the last month is measured on a 5 point scale, ranging from "never" to "very often". Higher scores reflect higher levels of perceived stress.
The change from baseline to endpoint in the Profile of Moods Scale-Brief Form (POMS-BF) | Baseline, Week 4
  The POMS-BF is a 30 item, self-report inventory in which a series of mood states (such as "Tense" or "Worn out") are rated based on how well each item describes the respondent's mood during the past week, including today. Items are rated on a 5-point scale with response options of: "Not at all", "A little", "Moderately", "Quite a bit" or "Extremely" with a global score range of 0 to 120 or individual domain scores on Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Lower scores indicate better mood state.
The change from baseline to endpoint on the Medical Outcomes Study- 12-item Sleep Scale Acute - Revised (MOS Sleep-R) | Baseline, Week 4
  The MOS Sleep-R is a self-reported scale containing 12 items addressing dimensions of sleep. It comprises six subscales: sleep disturbance, snoring, shortness of breath or headache, sleep adequacy, sleep somnolence, and sleep quantity. Items are answered on 5-point scales, where 1="all of the time," and 5="none of the time," 1 item (sleep latency) is answered on a 5 point scale from 1="0-15 minutes" to 5="more than 60 minutes." Score range of 0 to 100, where higher scores indicate fewer sleep-related problems. Duration of sleep is scored as the average number of hours slept per night.
The number of patients with a Hamilton Depression Rating Scale (HDRS17) anxiety/somatization factor score ≥7 at Week 4 | Week 4
  The HDRS17 is a clinician-administered rating scale designed to assess the severity of symptoms in patients diagnosed with depression with a score range of 0 to 52. Questions are related to symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss. The higher the score, the more severe the depression.
The number and percentage of patients with either ≥50% or ≥30% improvement on the HDRS17 total score at Week 4, and number and percentage of patients with HDRS 17 total score ≤ 7 at week 4 | Week 4
  The HDRS17 is a clinician-administered rating scale designed to assess the severity of symptoms in patients diagnosed with depression with a score range of 0 to 52. Questions are related to symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss. The higher the score, the more severe the depression.
The number of patients at Week 4 with ≥ 50% improvement on the SIGH-A (Structured Interview Guide of the Hamilton Anxiety Scale 14-item HAM-A) total score | Week 4
  The (HAM-A) is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. The answers range from 0 which signifies a complete lack of that symptom to 4, which indicates a very severe show of anxiety with that symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- Bulgaria (5):
  - Burgas
  - Kazanlak
  - Rousse
  - Sofia
  - Varna
- Hungary (4):
  - Baja
  - Budapest
  - Gyõr
  - Kalocsa
- Chisinau, Moldova
- Romania (2):
  - Arad
  - Iași
- Russia (5):
  - Nizny Novgorod
  - Saint Petersburg
  - Saratov
  - St-Peterburg
  - Tomsk
- Ukraine (9):
  - Donetsk
  - Hlevakha
  - Kharkiv
  - Kiev
  - Lviv
  - Odesa
  - Smila
  - Uzhhorod
  - Village Stepanovka Kherson